CLINICAL TRIAL: NCT04743102
Title: Study on the Value of Multi-points and Full-thickness Biopsy in the Diagnosis of Clinical Complete remiSsion After Neoadjuvant Therapy for Rectal Cancer
Brief Title: Multi-points and Full-thickness Biopsy in the Diagnosis of cCR After Neoadjuvant Therapy for Rectal Cancer
Acronym: BIOPSY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zhen Jun Wang, Professor, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIOPSY-01
Record Dates: First submitted 2021-02-04; First posted 2021-02-08 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Rectal Cancer; Neoadjuvant Therapy; Complete Remission; Metastasis
Keywords: rectal cancer; neoadjuvant therapy; clinical complete remission; full-thickness biopsy; watch-and wait; regrowth
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biopsy cCR (Experimental): Based on digital examination, serum CEA level, rectal MRI, endoscopy presentation, we add multi-points and full-thickness Biopsy to further improve the accuracy of cCR after neoadjuvant therapy for rectal cancer.
  Interventions: Procedure: multi-points and full-thickness Biopsy
- Conventional cCR (Active Comparator): Based on digital examination, serum CEA level, rectal MRI, endoscopy presentation, to study accuracy of cCR after neoadjuvant therapy for rectal cancer.
  Interventions: Diagnostic Test: traditional cCR

INTERVENTIONS:
Procedure: multi-points and full-thickness Biopsy — Four points around the tumor site and center of the tumor site full-thickness Biopsy
  Arms: Biopsy cCR
Diagnostic Test: traditional cCR — diginal examination, endoscopy test, rectal MRI, and serum CEA level
  Arms: Conventional cCR

SUMMARY:
Background There is currently no reliable means to restage rectal cancers after neoadjuvant chemoradiation. There are still no reliable methods to identify patients with pCR before radical surgery. As a result, clinical complete response (cCR), defined as no clinical detectable tumor by physical examination, endoscopic evaluation, and imaging, is designed as a surrogate endpoint for pCR. However, the concordance between cCR and pCR varies from 22% to 96% in different reports, which questions the clinical value of such strategies. Therefore, based on rectal diginal examination, serum CEA, MRI, endoscopy examination, we suggested to add multi-points and full-thickness biopsy technique to further improve the accuracy of cCR.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female, between 18 and 80 years old;
* Colonoscopy biopsy pathology confirmed colorectal adenocarcinoma;
* The distance from the lower margin of the tumor to the anal margin ≤12 cm (endoscope) or to the anorectal ring ≤8 cm;
* The hematopoietic functions of heart, lung, liver, kidney and bone marrow meet the requirements of surgery and anesthesia;
* Initial local MRI stage was T2 or T3A or T3B, N0-2, negative for extramural vascular invasion (EMVI), circumferential ential resection margin (CRM), and no peripheral iliac, common iliac, obturator, or abdominal aortic lymph node metastasis;
* CCR patients evaluated after neoadjuvant therapy (no mass or ulcer found on digital rectal examination;Endoscopic examination showed no other changes except flat scar, telangiectasia or pallor of mucosa.MRI or rectal ultrasound showed no residual tumor in the primary site and lymphatic drainage area.Serum carcinoembryonic antigen (CEA) was normal.
* Signing informed consent for surgery.

Exclusion Criteria:

* Previous history of malignant colorectal tumor;
* Patients complicated with intestinal obstruction, intestinal perforation, intestinal bleeding and other patients requiring emergency surgery;
* Unresectable lymph node metastasis;
* Recently diagnosed with other malignant tumors;
* Patients who had participated in or were participating in other clinical trials within 4 weeks prior to enrollment;
* ASA rating ≥IV and/or ECOG physical status score ≥2 points;
* Patients with severe liver and kidney function, cardiopulmonary function, coagulation dysfunction or combined with serious basic diseases cannot tolerate surgery;
* a history of serious mental illness;

  - pregnant or lactating women;
* Those with uncontrolled infection;
* Patients with other clinical or laboratory conditions considered by the investigator should not participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Complete Response rate | 8-12 weeks after preoperative chemoradiotherapy for locally advanced rectal cancer
  Clinical complete response rate between two groups after examinations following preoperative chemoradiotherapy for rectal cancer
pathological complete remission | 2 weeks after patients received radical operation
  No tumor cell found in surgical specimens

SECONDARY OUTCOMES:
Disease Free Survival | 5 years after operation or "watch and wait" approach
  no tumor regrowth or recurrence or metastasis found
Overall Survival | 5 years after operation or "watch and wait" approach
  survive during following

CONTACTS AND LOCATIONS:
Overall Officials: Zhenjun Wang, Study Chair — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No